CLINICAL TRIAL: NCT06819228
Title: Window Trial of Fluorescently Labeled Panitumumab (Panitumumab-IRDye800) in Head and Neck Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Eben Rosenthal, Barry and Amy Baker Professor and Chair, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: VICCHNP24602
Record Dates: First submitted 2025-01-24; First posted 2025-02-11 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: HNSCC; HNSCC,Larynx, Pharynx and Oral Cavity; SCC - Squamous Cell Carcinoma
Keywords: Pan800; Panitumumab; Fluorescent guided surgery; oral cancer; mouth cancer; tongue cancer; gum cancer; SCC; head and neck cancer; pharynx; HNSCC; larynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Laryngeal Diseases; Carcinoma, Squamous Cell; Mouth Neoplasms; Tongue Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1a - Cohort 1c (Experimental): These cohorts will receive one dose each of Pan800 (50 mg) and Panitumumab at a range of doses (varying of specific cohort).
  Interventions: Drug: Panitumumab IRDye 800
- Cohort 2a - Cohort 2c (Experimental): These cohorts will receive one dose of Pan800 and and two doses of Panitumumab at a range of doses (varying of specific cohort).
  Interventions: Drug: Panitumumab IRDye 800

INTERVENTIONS:
Drug: Panitumumab IRDye 800 — Study participation would last approximately 60 days from screening to follow-up visits. Participants dose of Panitumumab would be based on weight and Panitumumab IRDye800 is dosed the same for all participants.

SUMMARY:
This study is exploring the use of Panitumumab in Head and Neck Cancer. Panitumumab is an approved drug named Vectibix and is used as an anti-cancer agent in other cancers such as colorectal cancer. It works by attaching to the cancer cell in a unique way that allows the drug to get into the cancer tissue. In addition to the Panitumumab, participants will also receive a Panitumumab-IRDye800 (Pan800) or a fluorescently labeled Panitumumab infusion. IRDye800 is an investigational dye that, when tested in the lab, helps various characteristics of human tissue show up better when using a special camera during surgery. Panitumumab-IRDye800 is a combination of the drug and the dye that attaches to cancer cells and appears to make them visible to the doctor when he or she uses the special camera during surgery.

The goal of this study is to use a novel and possibly safer approach to identify an optimal dose for panitumumab to treat cancer patients by using a new light-based therapy. In this study, different drug levels will be analyzed using this approach to understand how much drug reaches the tumor at different administered doses, which may help us provide safer and/or more effective therapies in the future.

The goal is to identify the correct amount or dose of a drug that is needed for effective cancer therapies. Often, clinical studies look at how much of the drug can be tolerated before patients become sick, rather than how much of the drug is required to be effective.

IRDye800 is an investigational dye that, when tested in the lab, helps various characteristics of human tissue show up better when using a special camera during surgery. Panitumumab-IRDye800 is a combination of the drug and the dye that attaches to cancer cells and appears to make them visible to the doctor when he or she uses the special camera during surgery. This will help the surgeon with clinical margins during surgery and will may have a clearer way to differentiate between cancer and healthy tissue.

DETAILED DESCRIPTION:
The primary objective of this study is to understand biologic dosing of panitumumab which would contribute to the field by establishing new methodology for dose selection with the aim of reducing toxicity in cancer patients. For the individual patient in this trial, panitumumab itself is unlikely to demonstrate anti-tumor efficacy. However, previous studies have shown some benefit when using panitumumab-IRDye800 (pan800) as an imaging agent intraoperatively. The investigators hope to improve patient outcomes by gathering clinical data to support pan800 as a tool for reducing positive surgical margins and to identify malignant lymph nodes during surgical resection.

The drug being used in this study, panitumumab, is approved by the US FDA for treatment of certain types of advanced colorectal cancer at a dosage of 6 mg/kg given every 14 days. Many of the reported adverse events are associated with repeat administration of panitumumab, rather than 1-2 doses being administered in this study. However, the investigators do anticipate some adverse events at therapeutic dosing (anticipated grade 1-2). The most common side effects patients have experienced when receiving panitumumab primarily include skin reactions (including acne like rash, dry or itchy skin, cracking of skin around the participants nail beds, skin infections, and dry eyes), fatigue, nausea, and diarrhea.

Currently, there is no standardized method to identify the optimal biologic dose (OBD) for oncology therapies. Traditionally, dosing has been based on toxicity levels, specifically the maximally tolerated dose (MTD), rather than actual therapeutic effectiveness. In early-stage oncology trials, MTD often guides dose selection, with plasma drug concentrations serving as a rough measure for dose optimization. However, this plasma provides limited insight into how much of the drug actually reaches the tumor or binds to the intended target.

This study proposes a novel approach to finding OBD by measuring tumor drug concentration in head and neck cancer patients using an optically labeled antibody therapy. The investigators hypothesize that if a drug reaches a maximum concentration at a lower dose that previously thought, there may be no utility in increasing systemic dosing and risk unnecessary toxicity as well as financial burden.

Our group has previously published data using a fluorescent labeled therapeutic antibody (panitumumab-IRDye800) to show heterogenous distribution of antibody within a patient tumor in head and neck cancer. These studies used a single standard dose of panitumumab-IRDye800 which was shown to localize to malignant tumor tissue with minimal adverse events. In this proposed clinical trial, investigators will leverage this previously used fluorescent drug to investigate tumor concentration at multiple dose points up to and including the current FDA approved therapeutic dose to investigate our primary objective. Investigators will similarly use intraoperative fluorescence to assess the ability of the labeled antibody to distinguish malignant vs benign tissue at a range of doses. This intraoperative use has the potential to help optimize surgical margins and identification of malignant lymph nodes in addition to our primary objective of dose selection.

The main aim of this study is to investigate tumor concentration of fluorescently-labeled panitumumab at multiple doses up to the current FDA-approved therapeutic dose of panitumumab. This will allow us to identify if tumor saturation with this agent occurs below the currently approved dose. For other molecularly-targeted agents, there is evidence that lower doses can provide similar therapeutic benefit to approved doses. For panitumumab, over 30% of patients receiving this agent receive dose reductions due to adverse effects, resulting in a significant proportion of patients receiving a dose that is below the approved level. However, it is unclear if patients receiving this reduced dose achieve tumor saturation and similar therapeutic benefit. In this study, researchers will investigate if tumor saturation plateaus at a lower dose - an objective in line with dose optimization guidelines from the FDA. Our group has previously published data using fluorescently-labeled panitumumab to show heterogenous distribution of antibody within a patient tumor in head and neck cancer. Data from our previous and current work have allowed us to elucidate the relationship between fluorescence and intratumoral antibody concentration. An additional aim of this study is to provide further data on the efficacy of fluorescently-labelled panitumumab in identifying cancer relative to surrounding normal tissue. Improved tumor localization of the fluorescent agent could facilitate improved margin resections in the operating room.

ELIGIBILITY:
Inclusion Criteria:

* Willing to review and sign written informed consent.
* Male or female patients age > 18 years.
* Tissue confirmation of head and neck squamous cell carcinoma.
* Patients for whom a potentially curative resection is planned as standard of care.
* ECOG performance status of 0 or 1
* Adequate hematologic and end-organ function appropriate for surgery as determined by routine preoperative evaluation. If liver function, renal function and hematologic laboratory test results are acceptable for elective surgery, the patient is considered eligible for the study. Laboratory results that will need to be obtained within 30 days prior to initiation of study treatment: Magnesium, Phosphorus, serum pregnancy test (for females of childbearing age).
* For women of childbearing potential: Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods as defined below:

  • A woman is considered to be of childbearing potential if she is post-menarchal, has not reached a postmenopausal state (12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of the uterus and/or both ovaries and/or both fallopian tubes). Post-menarchal is defined as either:
  * age >55 years old
  * age <55 years or less and
* at least 12 months since last menstrual period,
* at least 6 months since last menstrual period and FSH > 40 IU

  * Women of childbearing potential must have a negative pregnancy test result within 14 days prior to initiation of study treatment.
  * Women must remain abstinent or use effective contraceptive methods during the treatment period and for 5 months after the final dose of panitumumab.
  * Men must agree to remain abstinent or use a condom during the treatment period and for 5 months after the final dose of panitumumab/pan800 to avoid exposing the embryo. Men must agree to refrain from donating sperm during this same period.

Exclusion Criteria:

* Patients not eligible for standard of care surgical resection
* Patients with a history of infusion reactions or allergic reactions to panitumumab.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.

  • History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Active tuberculosis. Patients do NOT have to be screened for tuberculosis for this trial.
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
* Patients receiving Class IA (quinidine, procainamide) or Class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents. The following drugs are known to interact with panitumumab and therefore any patients taking these medications within 30 days will be ineligible for the trial.
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of study treatment.
* Magnesium or phosphorus lower than normal institutional values, patient is symptomatic, and the values are unable to be corrected through standard repletion strategies.
* Evidence of QT prolongation on pretreatment ECG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Determine maximum tumor concentrating dose (MTC) of panitumumab in HNSCC. | Up to 21 days per patient
  Drug concentration in the tumor will be measured (drug ng/tissue mg) utilizing special imaging devices (such as the Tecan Spark, LI-COR Pearl Trilogy, LI-COR Elvis, and LI-COR Odyssey). These devices will only be used once the tissue is removed per Standard of Care during surgery and then comparing cancerous tissue to healthy tissue.
  The maximum tumor concentrating dose will be defined as the lower dose of drug after two consecutive doses demonstrate the same maximum concentration of intra-tumoral drug. The investigators will further evaluate if multiple doses are required to fully concentrate HNSCC in Cohort 2. The MTC dose with 1 vs 2 infusions preoperatively will be compared.

SECONDARY OUTCOMES:
Determine the efficacy of panitumumabIRDye800 to identify cancer compared to surrounding normal tissue | Up to 30 days per patient
  Tumor to background ratio (TBR) at various doses intraoperatively and on pathology. Pan800 fluorescence will be used to investigate image guided surgery with intraoperative imaging to optimize surgical resection. During the surgery, researchers and investigators will be able to utilize the PDE NIR Camera to visualize the Panitumumab IRDye800 during surgery. Investigators have used this for other studies with Panitumumab IRDye800, we do not anticipate this adding any additional risks to the patient. This will be utilized intraoperatively to evaluate correlation of fluorescence with clinical margins and postoperatively to correlate with tumor pathology in primary tumor specimens and metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: Eben L Rosenthal, MD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
This is a Pilot study at a single site in the U.S. The investigators do not plan to share IPD with other researchers at this time.

DOCUMENTS (1):
  • Informed Consent Form (2025-08-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT06819228/ICF_000.pdf